# <u>Strengthening Referral Networks for Management of Hypertension Across the Health System</u> (STRENGTHS): A Cluster Randomized Controlled Trial

# Dr. Constantine Akwanalo (Contact-PI)

Moi University College of Health Sciences and Moi Teaching and Referral Hospital 3-30100, Eldoret, Kenya

#### Dr. Jemima Kamano (MPI)

Moi University College of Health Sciences and Moi Teaching and Referral Hospital 3-30100, Eldoret, Kenya

# **Josephine Kisato (Project Coordinator)**

Academic Model Providing Access to Healthcare 4606-30100, Eldoret, Kenya

#### **Sponsor:**

The National Heart Lung and Blood Institute (NHLBI)

Grant Number: U01HL138636

Version: 9.0 – 2020-09-10 Version Date: 2020-09-10

# **Table of Contents**

| Lis | t of Tables | 4 |
|-----|---------------------------------------------------|----|
| Lis | t of Figures | 4 |
| Lis | t of Abbreviations | 4 |
| 1. | Synopsis | 0 |
| 2. | Study Flow | 1 |
| 3. | Background and Rationale | 2 |
| 4. | Specific Objectives | 2 |
| 5. | Concise Statement of Design | 3 |
| 6. | Participant Recruitment and Follow Up | 4 |
| I | nclusion Criteria | 4 |
| E | Exclusion Criteria | 4 |
| F | Recruitment Approach | 4 |
| F | Randomization | 4 |
| | Blinding | 5 |
| | Usual Care | 6 |
| | Intervention | 6 |
| F | Participant Follow Up | 7 |
| 5 | Study Withdrawal | 7 |
| 7. | Study Outcomes | 7 |
| ( | Clinical Efficacy Outcomes | 7 |
| F | Process Outcomes | 8 |
| ( | Cost Effectiveness Outcomes | 8 |
| 8. | Adverse Events and Serious Adverse Events | 8 |
| 9. | Data Collection, Handling and Record Keeping | 9 |
| | Data collection, handling and record keeping | 9 |
| F | Protections against risk to data | 10 |
| 10. | Data Analysis | 11 |
| N | Minimum detectable difference (MDD) | 12 |
| N | Methods of Analysis | 12 |
| F | Approach to handle missing data | 12 |
| 11. | Protection of human subjects | 13 |
| I | nformed Consent | 13 |
| | Data Safety and Monitoring Board | 13 |
| E | Ethical Approval | 16 |
| 12. | | |
| F | Policy on oral or written presentation of results | 17 |
| 13 | Timeline | 17 |

| 14. | References | 19 |
|---|---|---|
| 15. | Appendix | 23 |
| | Appendix 1: Screening for eligibility tool | |
| | Appendix 2: Consent Form STRENGTHS | |
| | Appendix 3: Process Evaluation Protocol | |
| | Appendix 4: Adverse Event and Serious Adverse Event Reporting Form | |
| | Appendix 5: Protocol Deviation/Violation Log | |
| | · | |

| <u>List of Tables</u> | |
|-------------------------------------------------------------------------|----|
| Table 1: Estimated power over a range of ICC and MDD values | 12 |
| Table 2: STRENGTHS Team Roster | |
| Table 3: Planned Enrollment by Sex | 18 |
| <u>List of Figures</u> | |
| Figure 1: STRENGTHS Study Flow | 1 |
| Figure 2: The Integrated HIT and Peer-support intervention | 3 |
| Figure 3: Referral Network Facilities in the STRENGTHS study | 5 |
| Figure 4: Adverse Events and Serious Adverse Events Reporting Procedure | |
| Figure 5: Timeline for overall STRENGTHS Study | |

# **List of Abbreviations**

| AE Adverse event | |
|---|---|
| AMPATH | Academic Model Providing Access to Healthcare |
| BP | Blood Pressure |
| CDM Chronic disease management | |
| VD Cardiovascular disease | |
| DALY | Disability-adjusted life year |
| DCC | Data coordinating centre |
| DSMB | Data Safety and Monitoring Board |
| EMR | Electronic medical record |
| ES | Executive secretary |
| FGD | Focus group discussions |
| HIT | Health Information Technology |
| ICC | Intra-class correlation |
| KII | Key informant interviews |
| LMICs | Low and middle-income countries |
| Lower-MICs | Lower middle-income countries |
| MDD | Minimum detectable differences |
| mHealth | Mobile Health |
| MTRH | Moi Teaching and Referral Hospital |
| NCD | Non-communicable disease |
| NHLBI | National Heart Lung and Blood Institute |
| PN | Peer navigator |
| RA | Research assistant |
| SAE Serious adverse event | |
| D Standard deviation | |
| SBP Systolic blood pressure | |
| SOP Standard operating procedure | |
| UC | Usual care |

# 1. Synopsis

| Title | Strengthening Referral Networks for Management of Hypertension Across the Health System (STRENGTHS) |
|---|---|
| Lead Institutions | Moi University College of Health Sciences (MUCHS) and Moi Teaching and Referral |
| | Hospital (MTRH) |
| Investigators | Dr. Constantine Akwanalo (MUCHS & MTRH) |
| | Dr. Jemima Kamano (MUCHS & MTRH) |
| | Dr. Benson Ng'ang'a (MTRH) |
| | Prof. Violet Naanyu (MUCHS) |
| | Dr. Ann Mwangi (MUCHS) |
| | Dr. Timothy Mercer (University of Texas, Austin) |
| | Dr. Rajesh Vedanthan (New York University) |
| | Dr. Sonak Pastakia (Purdue University) |
| | Dr. Jonathan Dick (Indiana University) |
| | Dr. Makeda Williams (NHLBI) |
| Study Sites | Primary, Secondary & Tertiary Health Facilities in Uasin Gishu County, Trans Nzoia |
| Study Citos | County, Busia County, Bungoma County and Nandi County |
| | Sounty, Busia Sounty, Bungoina Sounty and Nanai Sounty |
| Planned Study | 2017 - 2022 |
| Period | |
| Objective | This study aims to evaluate whether an integrated intervention composed of peer |
| | support and a health information technology tool can improve referral adherence and |
| | improve blood pressure among patients with complicated hypertension in a lower |
| | middle-income country setting |
| Study Design | This is a cluster randomized controlled trial that will compare: |
| | Intervention: An integrated intervention composed of peer support and a health |
| | information technology tool to support referral services |
| | Control: Usual referral service |
| | A total of 8 clusters representing unique referral networks will be randomized equally |
| | at the level of the secondary health facility. |
| Number of | 1600 patients with hypertension who are referred either to a higher or lower health |
| Participants | facility |
| Inclusion Criteria | Age ≥ 18 years and either: |
| | Patients with complicated hypertension (meet criteria for referral up the |
| | network), defined as any of: |
| | a. Uncontrolled (SBP ≥ 140 or DBP ≥ 90) on 3 or more anti-hypertensive |
| | medications |
| | b. Have signs or symptoms of end-organ damage (dyspnea on exertion, |
| | leg edema, reduced urine output, focal weakness) |
| | c. Have suspected secondary causes of hypertension (age <35 years, |
| | HIV, or pregnancy) |
| | d. Any other concerning condition that the clinician suspects to be |
| | attributable to hypertension for which they would seek a higher level of |
| | care |
| | Laic |

| | Or: |
|---|---|
| | <ol> <li>Patients with stable, uncomplicated hypertension (meet criteria for referral<br/>down the network), defined as controlled BP (SBP &lt; 140 and DBP &lt; 90) for 3<br/>or more consecutive visits and no evidence of new end-organ damage</li> </ol> |
| Exclusion Criteria | Acute illness requiring immediate medical attention |
| | 2. Terminal illness |
| | History of coronary artery disease or stroke |
| | Inability to provide informed consent |
| Primary Endpoint | One-year absolute mean change in SBP |
| Secondary | One-year change in overall CVD risk as measured by the QRISK2 score |
| Endpoints | Process Metrics |
| | Up-referral completion rate |
| | Down-referral completion rate |
| | Median referral completion time |
| | Referral appropriateness |

# 2. Study Flow



Figure 1: STRENGTHS Study Flow

# 3. Background and Rationale

**Hypertension: Burden and Implementation Gaps.** Elevated blood pressure (BP) is the leading preventable cause of early death and disability globally, <sup>1,2</sup> and 75% of patients with hypertension live in LMICs.<sup>3</sup> In Kenya, prevalence of hypertension is nearly 25%.<sup>4</sup> similar to. Despite many evidence-based interventions to manage hypertension, gaps in implementation persist, especially in LMICs.<sup>3,5,6</sup> In lower-MICs, only 37% of known hypertensives were on treatment, with less than 10% of them being adequately controlled.<sup>5</sup>\_

Referral Networks. The Kenya Health Referral Strategy 2014-2018 highlights an effective referral system as crucial to improving equitable access to essential health services. However, referral networks in Kenya and similar lower-MICs are characterized by referral non-adherence and delays in referral completion. Public sector health systems in lower-MICs often employ a multi-level system spanning a primary- to specialty-care continuum, with a tripartite system of primary, secondary, and tertiary care. Patients with complicated hypertension require referral up the network for specialty care, as well as advanced diagnostic and treatment modalities. Patients with stable, uncomplicated hypertension can be referred down the network where care is geographically decentralized and task-shifted to lower levels of providers, reducing costs and increasing access to care. Effective referral networks have improved outcomes in maternal and child health, HIV, 15,16 and CVD. Truthermore, in resource-limited settings, strong referral networks are essential to improve the efficiency of resource utilization and guarantee equitable provision of healthcare services. Therefore, strong referral networks provide an evidenced-based foundation upon which interventions for hypertension can be implemented and evaluated in lower-MICs.

Multi-Level Factors Impacting Referral Networks for Hypertension. Rates of referral adherence in lower-MICs is low. Successful referral completion was only 37% among patients found to have hypertension or at elevated CVD risk following community-based screening in Bangladesh, Guatemala, Mexico and South Africa. The Burkina Faso, referral adherence was 20% among patients referred for hypertension. The causes of referral non-adherence are multifactorial. The Patient-related factors include lack of time, cost, transport distances, and limited understanding of the rationale. Provider-level factors include poor documentation and limited human resources for health. Health system-related factors include lack of integrated health records, 23,24 long patient waiting times, and the complexity of navigating larger health facilities.

<u>Peer Support.</u> Peer-based care approaches leverage unique patient-patient interactions built on shared disease experiences to influence behavior change.<sup>25</sup> Peers have successfully been used to improve adherence to HIV medicines <sup>26-29</sup> and have effectively supported chronic disease management.<sup>7,30-33</sup> Peer navigators have been used to improve linkage to and retention in care for patients with HIV,<sup>34,35</sup> as well as improve healthcare utilization in mental health<sup>36</sup> and cancer.<sup>37,38</sup> To date, peer navigators have not been evaluated in the context of strengthening referral networks to improve hypertension control.

<u>HIT.</u> HIT, including integrated EMRs and mHealth, are a key strategy in LMICs for NCD management, <sup>39-41</sup> and can improve documentation and data capture, which are significant barriers to effective referral networks. <sup>13,23,42</sup> Our systematic review of mHealth for NCDs in sub-Saharan Africa highlights the use of HIT for patient follow-up and peer networks among patients with NCDs. <sup>43</sup> However, the evidence base is limited, with an urgent need for more rigorous implementation research of HIT interventions. <sup>43</sup> Specifically, it is not well known if HIT, in combination with peer support, can strengthen referral networks for hypertension control.

# 4. Specific Objectives

The objective of this research is to utilize the PRECEDE-PROCEED framework to conduct transdisciplinary, translational implementation research focused on strengthening referral networks for hypertension control. The central hypothesis is that HIT integrated with peer support will be effective and cost-effective in strengthening referral networks, improving BP control, and reducing CVD risk among patients with hypertension in western Kenya. We hypothesize that HIT and peer support will synergistically address barriers to hypertension control at the patient, provider and health system levels. We further hypothesize that changes in referral network\_characteristics may mediate the impact of the intervention on the primary outcome, and that baseline referral network characteristics may moderate the impact of the intervention. To test these hypotheses and achieve the

overall objective, we will conduct a two-arm cluster randomized trial comparing: 1) usual care vs. 2) referral networks strengthened with an integrated HIT and peer support intervention. We will pursue the following specific objectives:

- 1. Evaluate the effectiveness of HIT and peer support on one-year change in SBP and CVD risk reduction.
- 2. Conduct mediation analysis to evaluate the influence of changes in referral network characteristics on intervention outcomes, and a moderation analysis to evaluate the influence of baseline referral network characteristics on the effectiveness of the intervention.
- 3. Conduct a process evaluation using the Saunders framework, evaluating key implementation measures related to fidelity, dose delivered, dose received, recruitment, reach, and context.
- 4. Evaluate the incremental cost-effectiveness of the intervention, in terms of costs per unit decrease in SBP, per percent change in CVD risk score, and per DALY saved.

#### 5. Concise Statement of Design

We will evaluate the effectiveness of HIT and peer support for strengthening referral networks for hypertension control by conducting a non-blinded two-arm cluster randomized trial comparing: 1) usual care vs. 2) referral networks strengthened with an integrated HIT and peer support intervention (Figure 2). The primary outcome measure will be one-year change in systolic blood pressure (SBP) and a key secondary outcome will be change in CVD risk score.



Figure 2: The Integrated HIT and Peer-support intervention

# 6. Participant Recruitment and Follow Up

#### **Inclusion Criteria**

Adult patients (≥18 years) who are enrolled in AMPATH's CDM program with hypertension, who meet criteria for referral up or down the network, will be eligible for inclusion in the trial.

For referral up, criteria are:

- Patients with complicated hypertension, defined as any of:
  - a. Uncontrolled (SBP ≥ 140 or DBP ≥ 90) on 3 or more anti-hypertensive medications
  - b. Have signs or symptoms of end-organ damage (dyspnea on exertion, leg edema, reduced urine output, focal weakness)
  - c. Have suspected secondary causes of hypertension (age <35 years, HIV, or pregnancy)
- Any other concerning condition that the clinician suspects to be attributable to hypertension for which they would seek a higher level of care

For referral down, criteria is patients with stable, uncomplicated hypertension, defined as controlled BP (SBP < 140 and DBP < 90) for 3 or more consecutive visits **and** no evidence of new end-organ damage

#### **Exclusion Criteria**

- Acute illness requiring immediate medical attention
- Terminal illness
- History of coronary artery disease or stroke
- Inability to provide informed consent

### **Recruitment Approach**

The clinicians will be sensitized about the study and the eligibility criteria. They will then invite AMPATH CDM patients with hypertension and eligible for referral from the health facility to enroll in the study on the day of their routine clinic visit. On that day, research team members will briefly describe the research study to the potential participant. They will then perform a short interview using the screening for eligibility tool which documents the age of patient, type of referral and reason for referral (Appendix 1). Patients meeting eligibility criteria will then be asked their willingness to participate in the study, and if willing will proceed to the informed consenting stage. Patients not meeting eligibility or unwilling to participate further will be referred back to their clinician to continue with clinical care as per the clinician's management plan. For referral networks randomized to the HIT and peer support intervention arm, participants will be informed of the HIT functionality and the availability of peer navigators who can assist them with the referral process. Extreme care will be taken to fully explain the benefits and risks of the research study, before written consent is obtained. The consent will be written in lay terminology at approximately 6th grade (USA) level (Appendix 2). Individuals will be free to refuse to participate in the study at any time during the period of the study. A refusal will not impact the health care available to the individual in any manner. Access to care will not be impacted in any manner by an individual's decision to opt out of this research project.

#### Randomization

The unit of randomization will be a cluster, which consists of a geographically separate, distinct hypertension referral network within the overall AMPATH CDM program. There will be a total of eight clusters (referral networks), each of which will be centered around a secondary-level health facility: Mosoriot, Kwanza, Kiminini, Webuye, Kocholya, Bunyala, Butula, and Nambale (Figure 3). Each of these secondary-level facilities constitute the last step in their respective referral network before reaching the common, tertiary level of MTRH, Busia County Referral Hospital, Kitale County Referral Hospital, or Bungoma County Referral Hospital. In addition, each secondary-level facility has a number of primary-level health facilities that feed into it. Four of

the clusters will be randomly assigned to the intervention arm, and four will be randomly assigned to the control arm. Randomization will be stratified by the size of the secondary-level health facility.

| Clusters* | Primary Level | Secondary Level | Tertiary Level |
|---|---|---|---|
| Mosoriot | Mogoget<br>Birbiriet<br>Itigo<br>Lelmokwo<br>Kokwet<br>Ngechek | Mosoriot Sub-county hospital | Moi Teaching and<br>Referral Hospital |
| Kiminini | Bikele<br>Sister Fredah | Matunda Sub-county hospital | Kitale County |
| Kwanza | Kaisagat<br>Namanjala | Kwanza Sub-county hospital | Referral Hospital |
| Webuye | Milo | Webuye County hospital | Bungoma County |
| Kocholya | Angurai<br>Changara<br>Malaba<br>Kamolo<br>Akichelesit<br>Aboloi<br>Moding | Kocholya Sub-<br>county hospital | Referral Hospital |
| Bunyala | Budalangi<br>Bulwani<br>Busagwa<br>Mukhobola<br>Osieko<br>Rukala<br>Sirimba<br>Sisenye | Port Victoria Sub-<br>county hospital | Busia County<br>Referral Hospital |
| Butula | Bumala A<br>Bumala B<br>Ikonzo<br>Sikarira | Khunyangu Sub-<br>county hospital | |
| Nambale | Lwanyange<br>Madende<br>Musokoto | Nambale Sub-<br>county hospital | |

Figure 3: Referral Network Facilities in the STRENGTHS study

#### **Blindina**

Trial participants, research assistants and the research coordinator will not be blinded. This is because the nature of the intervention, peer support, cannot be concealed from participants, or the research staff who will be doing enrollment and follow-up at the clinic sites and as such will be aware if there is a peer or not in the facility. The data analyst/biostatistician and co-investigators will be blinded, unaware which participant is assigned to which arm of the trial. The Pl's (CA and JK) see patients at the cardiology and medical outpatient clinic at MTRH, and might interact with study participants during their clinical duties. They might therefore become aware, during the course of their clinical duties, of the trial arm to which a study participant has been

<sup>\*</sup>Unit of randomization

assigned. Should this happen, the PIs are expected to implement usual clinical care regardless of the patient's participation in the trial. No further action will require to be taken.

#### **Usual Care**

Within the AMPATH CDM program, usual management at the primary and secondary levels involves an attempt to control BP with up to 3 anti-hypertensive medications before referral, under the supervision of a mentoring clinician who visits the lower level facility on a rotating basis. Frequency of clinical visits will depend on clinical circumstances and level of care, mimicking real-word conditions. The process for referrals will continue as it is currently practiced within the AMPATH CDM program and Kenyan MOH. For patients with complicated hypertension requiring referral up the network, the referring clinician writes a referral letter on a standardized, blank referral form, with demographic information of the patient and reason for referral. This referral letter is then given to the patient, who is responsible for presenting it to the receiving facility and arranging the referral visit. For patients with stable, uncomplicated hypertension requiring referral down the network, a counter-referral letter, and/or copies of clinical records, are given to the patient to take back to their primary facility, although this process is not consistently adhered to. There is no dedicated psychosocial or health system navigation support in the usual care arm.

#### Intervention

Those randomized to the intervention group will receive clinical care for hypertension in the same manner as those randomized to the usual care group. Reasons for referral will also be the same in the two groups. The change in referral process is the intervention which is an integrated HIT tool and peer support.

<u>HIT</u>: AMPATH uses AMRS, a customized version of OpenMRS.<sup>44</sup> AMRS is centrally hosted and accessed by tablet via the Internet with all data simultaneously available to all users of the system, independent of their location. This facilitates both real-time data collection and monitoring. Our HIT intervention will augment AMRS to support a referral system in four ways: 1) <u>communication</u>: facilitate data sharing by all providers and peer navigators across all levels of the health system; 2) <u>decision support</u>: provide clinical decision support to facilitate appropriate patient referrals; 3) <u>tracking</u>: generation and sharing of real-time patient referral lists; and 4) <u>dashboards</u>: create a platform for monitoring key evaluation metrics. The system will prompt for referral if indicated but also allow the user to self-initiate a referral. Providers and peer-navigators will access the designed referral dashboard for a clinic to review patient referrals, identify patients who made their referral appointment, and track patients who have been referred back to the referring site. Key referral process metrics (described below under "Secondary Outcomes") will be available in real-time for providers and peer navigators to monitor and act upon.

Peer Support: The peer support component of the intervention will involve "peer navigators" at each level of the referral network – primary, secondary and tertiary, titled "Community Peer Navigators", "Facility Peer Navigators", and "Central Peer Navigators", respectively. The Community Peer Navigators will cover a catchment area within the community surrounding each primary level health facility. The Facility Peer Navigators will be stationed at the secondary level health facilities in each referral network. The Central Peer Navigator will be stationed at the tertiary level, MTRH. The roles of the peer navigators will be drawn from those described in the HIV and oncology literature, 45-50 but adapted and contextualized. The peer support intervention has three main functions: 1) referral adherence: link clinicians and patients to provide referral logistics support; 2) <u>navigation</u>: help patients navigate the complex health system;<sup>51</sup> and 3) <u>psychosocial</u> support: leverage their shared disease experience to help patients overcome barriers to health seeking behavior. Referral adherence support entails ensuring patients know the "what, where, when, and how" of the referral process. The peer navigators will be equipped with an HIT tool, as described above, so they can see the same data as the clinicians in order to track and follow referred patients appropriately. When a clinician at the primary level refers a patient to a higher level of care, the Community Peer Navigator covering that patient's community catchment area will automatically be alerted on their HIT tool so they can contact and meet the patient, and review referral logistics. The Community Peer Navigator will then complete a referral navigation form on the HIT tool, which will automatically trigger a notification to the clinician and Facility or Central Peer Navigator at the receiving facility, alerting them of the incoming referral. The second major role of the peer navigator is health system navigation, especially at the tertiary level. Here, the peer navigator can

personally and physically receive a referred patient and walk them through the complexities of registration, scheduling, triage, and diagnostic work-up in order to streamline the referral process and ensure patients are not lost in the complexity of the system.<sup>52</sup> Furthermore, peer navigators will meet with patients after the clinic visit to provide any follow-up navigation between the pharmacy, laboratory, or imaging. Communication between the Central, Facility, and Community Peer Navigators will be automated via the HIT tool to ensure seamless communication and data-sharing. The third major role of the peer navigator is to provide psychosocial support to patients and their families, helping them overcome individual-level barriers to health seeking behaviors, drawing from the innate trust inherent in their shared disease experience.<sup>25</sup> Peer navigators at all levels will be trained to provide education, motivational interviewing, and psychosocial support.

#### **Participant Follow Up**

Participants will have three visits for both study arms: a baseline visit upon enrollment, a six-month visit, and a 12-month visit. In both arms of the trial, if the patient does not present to the clinic for the 6 month or 12-month visit, the patient will be traced by the research team. Missing data resulting from loss to follow up will be handled as detailed in section 10.

#### Study Withdrawal

Individuals will be free to refuse to participate in the study and withdraw at any time during the period of the study. Withdrawal will not impact the health care available to the individual in any manner. Access to care will not be impacted in any manner by an individual's decision to opt out of this research.

#### 7. Study Outcomes

#### **Clinical Efficacy Outcomes**

# **Primary outcome**

#### One year absolute change in mean BP

The systolic blood pressure at baseline will be compared to systolic blood pressure after 1 year of follow up.

#### **Secondary outcomes**

#### One-year change in overall CVD risk as measured by the QRISK2 score

QRISK2 score is a computerized algorithm for predicting the ten-year risk of developing CVD events. The factors that enter into the calculation of the QRISK2 score include: Age 25-84 years, sex, ethnicity, smoking status, diabetes status, family history of coronary artery disease in first degree relatives below the age of 65 years, chronic kidney disease stages 4 and 5, atrial fibrillation, rheumatoid arthritis, cholesterol / high density lipoprotein ratio, systolic blood pressure, body mass index.

A score of 10% or more suggest a 10% risk of primary CVD events in ten years and warrants intervention to reduce the risk. It's not used among patients who already have a heart attack or a stroke.

#### One-year mortality rate

Death by the end of the 1 year follow-up

#### **Hospital admissions**

Number of self-reported hospital admissions for any cause among participants over one year follow up

#### CVD complications

Any self-reported cardiovascular complications including hypertensive crises, heart failure, Stroke and Acute myocardial infarction

#### Change in CVD risk factors and behaviors

Baseline risk factor profile compared to profile at 1 year of the various CVD risk factors as assessed using a standardized CVD risk factors and behaviors screening questionnaire

#### **Medication adherence**

Changes in self-reported adherence to hypertension medication at one year from baseline as assessed using the Voils adherence questionnaire<sup>53</sup>

#### **Process Outcomes**

Referral Process Metrics

- Up-referral completion rate
- Down-referral completion rate
- Median referral completion time

#### **Process Evaluation**

- Fidelity (quality of intervention delivery as assessed using a checklist-based field observation of peer navigators, written tests for peer navigators at baseline and six months, and separate focus group discussions for peer navigators, participants and clinicians, see Appendix 3 for full Process evaluation protocol)
- Dose delivered (completeness)
- Dose received (exposure and satisfaction)
- Recruitment
- Reach (participation rate)
- Context

#### **Cost Effectiveness Outcomes**

Incremental cost effectiveness ratio

#### 8. Adverse Events and Serious Adverse Events

An AE is defined as any untoward or unfavourable medical occurrence in a human subject, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the subject's participation in the research, whether or not considered related to the subject's participation in the research.

### An SAE is a defined as any AE that:

- results in death;
- is life-threatening (places the subject at immediate risk of death from the event as it occurred);
- results in inpatient hospitalization or prolongation of existing hospitalization;
- results in a persistent or significant disability/incapacity;
- results in a congenital anomaly/birth defect; or
- based upon appropriate medical judgment, may jeopardize the subject's health and may require medical or surgical intervention to prevent one of the other outcomes listed in this definition

The safety observation period extends from the time the signed informed consent is obtained through the completion of the final study visit. All patients enrolled in the trial who experience an SAE will be managed at their nearest health facility according to the Kenya MOH cardiovascular disease guidelines,<sup>54</sup> with referral to higher levels of care if needed.

#### **Reporting Procedures**

Given that peer navigators and research assistants are the study staff who will have direct contact with study participants, we anticipate that an AE or SAE will first be detected by the peer navigator or the research assistant. Should the PN be the first to detect a probable AE or SAE, they will be expected to report to the RA within 1 hour of detection. Once an RA is aware of an AE or SAE, they will fill out the electronic AE/SAE reporting form (Appendix 4), and inform the research coordinator via phone, both RA actions will be expected to be complete within 1 hour. The filed form will then be reviewed by one of the three clinical Kenyan investigators within four hours, who will then ascertain the AE/SAE. If ascertained as a true AE/SAE, the investigator will be expected to generate a report to NHLBI, IREC and the DSMB within 24 hours. All peer navigators and RAs will be trained on AEs and SAEs detection and reporting. All SAEs and AEs will be captured on electronic CRF. The three Kenyan clinical investigators (a monthly rota will be created and maintained by the research coordinator) are responsible for continuing to follow all AE and SAE reports (whether or not related to study intervention) until resolution or until the event is considered chronic and/or stable by the investigator and/or other physician who has the responsibility for the patient's medical care. All SAEs will require expedited reporting by the PI to the study's DSMB, IREC/IRB, and NHLBI. An expedited report of an SAE will be submitted by email and must be reported to the DSMB, IREC/IRB and the NHLBI within 24 hours of the event being reported to the Investigator. The expedited report will be followed by a detailed, written AE/SAE report using the standard study AE/SAE reporting form (Appendix 4) as soon as possible. Follow up information will be availed if asked for by DSMB directly, or from NHLBI or its representatives. A master log of all AE's/SAE's will be maintained and the PI will submit a statistical report from the log to the DSMB at least two weeks prior to all scheduled DSMB meetings.



Figure 4: Adverse Events and Serious Adverse Events Reporting Procedure

# 9. Data Collection, Handling and Record Keeping

#### Data collection, handling and record keeping

For the primary and secondary clinical efficacy outcome, the baseline and 12-month assessments will be measured by trained study staff to ensure standardization and uniformity of measurement. Data will be collected on covariates we hypothesize may be related to our outcomes. These include patient demographics, socioeconomic and education status, clinical comorbidities, CVD risk factors, health behaviors, geographic location, referral level, and provider level of training.

For the process outcomes, data will be collected at whatever level of care the patient clinically requires, in order to mimic real-world practice and accurately map the patient wherever he or she falls within the referral network. Semi-quantitative and qualitative data for the process evaluation, including observation, surveys, interviews, and focus group discussions. Observational data will not contain any patient identifiers. These data include transcripts of mabaraza<sup>55</sup> (traditional form of community assembly), focus group discussions, and interviews; completed clinician surveys; and observation notes (study activities preceding the trial portion). Mabaraza, focus group discussions, and interviews will be digitally audio-recorded and uploaded with a coded identification number (no identifying names) as an audio file to an electronically secure database. Similarly, the clinician surveys will be de-identified and coded, and the data extracted and stored in the same electronically secure database. These research data will be stored in an electronically secure database protected by password that will be known only to key research team members and the Study Coordinator. Once uploaded to the electronically secure database, the data will be deleted from the digital recording device and the original surveys containing identifying information will be destroyed. Electronically captured data will transfer to the research database at the time of entry into the handheld device through a secure connection tunnel. All data on mobile devices will be encrypted and stored on the device's internal memory. All paper data collection forms will be reviewed by the Study Coordinator and Data Manager for completeness. Once validated, any sheets containing directly identifiable information and consent documentation will be separated and added to the site's secure storage locker. The remaining, de-identified pages will then be placed in a separate storage locker prior to data entry. Only key investigators and study personnel will have access to individually identifiable private information about human subjects. Transcription of the audio files will occur in Kenya and will be done by the trained research assistants. These transcripts will also be stored in an electronically secure database on a password-protected computer.

For the cost-effectiveness outcomes, cost data will be obtained during the implementation of the intervention and health service utilization data will be obtained from the AMRS. These data will be collected during the course of the project implementation by research staff. Two sets of costing instruments will be used, one completed by study participants, and the other completed by research staff. The instruments completed by participants capture healthcare utilization and expenditures, work loss, and transportation costs and can be used to quantify cost offsets from intervention participation. The instruments completed by research staff capture all relevant labor, materials, supplies, and contracted services costs for all activities required to deliver the intervention. All data collected on paper forms will be transferred to the research database using double data entry.

Electronically captured data on REDCAP will transfer to the research database at the time of entry into the handheld device through a secure connection tunnel. All data on mobile devices will be encrypted and stored on the device's internal memory. All paper data collection forms will be reviewed by the Study Coordinator and Data Manager for completeness and the presence of pre-specified "danger" values. Once validated, any sheets containing directly identifiable information and consent documentation will be separated and added to

the site's secure storage locker. The remaining, de-identified pages will then be placed in a separate storage locker prior to data entry. Only key investigators and study personnel will have access to individually identifiable private information about human subjects.

#### Protections against risk to data

The following principles and procedures for data collection will be followed at the research site in order to minimize risk and protect confidentiality:

- Data will be collected on coded forms, which do not include other personal identifiers
- Only the tracking form will have the participant's name and identifiable information
- Study records will be stored in locked cabinets in a locked room
- Only the study personnel will have access to the data and the codes
- All computerized information will be protected by access codes known only to key investigators and certain designated staff members
- No data will be published with participant names
- Data that are contained on a digital audio recording device will be PGP-encrypted
- All staff members will be trained to keep participants' information confidential, and will be informed of the penalty for breach of confidentiality

The consent form signed by the participant will provide written assurance that all individual data collected in the study will be kept confidential to the extent provided by the Privacy Act of 1974. AMPATH will provide file security so that confidential data are not released. Specifically, participants will be informed that: (1) the only people who will know that they are research participants are members of the research team and, if appropriate, their physicians or health care providers; (2) no individual identifying information about them will be disclosed to others, except if required by law; and (3) when the results of the study are published or discussed in conferences, no information will be included that would reveal their identity.

Any material that is digitally audio-recorded will be uploaded with a coded identification number (no identifying names) as an audio file to an electronically secure database. These research data will be stored in an electronically secure database protected by password that will be known only to the Principal Investigator and the Study Coordinator. Once uploaded to the electronically secure database, the data will be deleted from the digital recording device. Transcription of the audio files will occur in Kenya. These files will also be stored in an electronically secure database on a password-protected computer.

All clinical patient-level data will be entered into the AMRS as per AMPATH's standard operating procedures. A separate, password-protected research database will retrieve data from AMRS via access that will be controlled through user authentication. All data collected on paper forms will be transferred to the research database using double data entry. Electronically captured data will transfer to the research database at the time of entry into the handheld device through a secure connection tunnel. All data on mobile devices will be encrypted and stored on the device's internal memory.

All data management will be carried out by CITI-certified research staff members, and all data will be stored on dedicated, password-protected computers. Any data stored on portable media will be PGP-encrypted, in order to ensure security of the data. Paper forms will be stored for the duration of the study, and for one year following in order to allow verification of any data as needed for reporting and publication purposes. The paper forms will then be shredded. The electronic data with a coded identification number only (and no identifying names) may be kept indefinitely, in a secure manner as described above.

To prevent inadvertent disclosures and ensure subject confidentiality, data entry and document storage for materials containing directly identifiable information (i.e., coversheets) will be handled by key investigators or the Study Coordinator. The Study Coordinator will be responsible for the secure handling and storage of survey documents for the duration of research activity at the study site. Once activities have been completed, coversheets will be collected and forwarded to the AMPATH research office, where they will be stored in a secure, locked cabinet within a secure, locked room. To minimize the number of people with access to the

coversheet data, all data entry will be conducted under the direct supervision of the Study Coordinator. Once identifiable data has been entered as described, paper-based documents will be returned to secure storage.

#### 10. Data Analysis

We will quantify the effectiveness of an integrated HIT and peer support intervention for strengthening referral networks to improve BP control and reduce CVD risk. The primary outcome measure is one-year absolute mean change in SBP. A key secondary outcome measure is one-year change in overall CVD risk as measured by the QRISK2 score, which has been validated for calculating 10-year CVD event risk for Black Africans. 146-154

For the cost-effectiveness analysis, only net incremental costs, after factoring in cost offsets that may result from improved health, will be included as the numerator in the CE analysis as these are the relevant costs for decision makers. As part of the costing analysis, we will also identify which activities drive the overall costs, and how costs would change if specific activities are added or eliminated.

#### Minimum detectable difference (MDD)

The study is powered to detect improvement in SBP in the intervention arm compared to usual care. We expect that each of the eight referral networks will enroll at least 200 participants. Based on other studies in the region we expect a difference of 4 to 10-mmHg<sup>56</sup> between the two groups at month 12. The power calculations summarize MDD in the primary outcome for the comparison between the two groups. Using a two sided test with a Type I error rate at 5% (alpha = 0.05), and a standard deviation of 15mmHg (SD values for change in SBP found in the literature ranges from 10 to 20). Table 1 presents power for the comparison across different combinations of ICC ranging from 0.02 to 0.08, consistent with prior studies using SBP as the outcome Table 10 mmHg. We assume that up to 15% of enrolled participants will be lost to follow up.

Table 1: Estimated power over a range of ICC and MDD values

| | ICC | | | |
|-----|------|------|------|------|
| MDD | 0.02 | 0.04 | 0.06 | 0.08 |
| 4 | 52 | 32 | 24 | 20 |
| 6 | 85 | 61 | 46 | 37 |
| 8 | 98 | 84 | 70 | 58 |
| 10 | 99 | 96 | 87 | 77 |

#### **Methods of Analysis**

Our analyses for both the primary and secondary outcome will be conducted according to the principle of intention to treat, in which every cluster is analyzed according to the assigned intervention, regardless of the treatment actually received. We will use a repeated measures mixed-effects model for SBP, with fixed effects for time and intervention arm, and random effects for cluster and individual. The model specification is:

$$E\big(Y_{\mathit{itk}}\big) = \alpha + \beta_1 I\big(t = 6\big) + \beta_2 I\big(t = 12\big) + \beta_3 I\big(t = 6\,, intervention\big) + \beta_4 I\big(t = 12\,, intervention\big)$$

where  $Y_{itk}$  is SBP for the  $i^{th}$  individual at the  $t^{th}$  time in the kth cluster and I() represents the indicator of the event in (). The hypothesis test for the coefficient  $\beta_4$  will be a test of whether SBP after 1 year differs for those in the intervention compared to those in the usual care condition.

We will compare key independent variables across the trial arms to ensure balance of the randomization process, and assess whether adjustments for any baseline characteristics is necessary and make adjustments in the model to estimate treatment effects as needed. The analysis will be stratified by predefined strata of referral up and referral down. For modeling QRISK2, we will use the transformation log (log(QRISK2)) because the risk score ranges from 0% to 100%. The model will be fit using maximum likelihood with the software package R.

# Approach to handle missing data

Individuals who are missing outcome data at 12 months will be traced by the research team to ascertain and alleviate dropout bias in our trial. The follow-up sample will enable us to form an imputation model for the missing outcomes. Using the subset of individuals who dropped out but whose SBP was ascertained after tracing, we will fit a regression using 12-month outcome as the dependent variable, and baseline covariates and the most recently observed outcome at month 6 as the independent variables, and use the model to generate predicted (imputed) values of outcomes for those not traced. We will account for uncertainty using multiple imputation. In addition, the generalized linear mixed models proposed for the primary and secondary analyses incorporate an assumption of data that are missing at random, meaning that the likelihood of a value being missing depends on observable characteristics. We will employ sensitivity analyses via pattern mixture modeling participants (expected to be up to 15% of the sample, as above).

#### 11. Protection of human subjects

#### **Informed Consent**

The proposed study will be conducted following strict guidelines for the protection of the rights of participants. Informed consent will be signed by all participants following screening. Extreme care will be taken to fully explain the benefits and risks of the research study, before consent is obtained. Written informed consent will be obtained from all participants. The consent form (Appendix 2) will be written in lay terminology at approximately 6th grade level. Participation in the study will be discontinued if the participant chooses to stop participating in the study and notifies the study team. Participants will be allowed to withdraw from the study, should they choose to, without risk of any discrimination, or any risk of impact on their clinical care and they can choose to seek clinical care at any facility (AMPATH, other public sector or private sector) that they wish.

The residents of study site areas may come from economically disadvantaged backgrounds. We will continue the policy of AMPATH of not providing excessive monetary compensation for study subjects beyond reimbursement to cover travel expenses and time. This policy will be followed in order to ensure that consent is freely given without risk of "monetary coercion." Vulnerable populations such as children, neonates, human fetuses, and any individuals <18 years old will not be included in the study. Pregnant women who are hypertensive will be eligible for participation in the trial but their clinical management will remain per the usual clinical care. Within each referral network cluster, the relevant MOH facilities will be contacted and receive information on the different study procedures anticipated through completion of this project.

# **Data Safety and Monitoring Board**

An independent DSMB has been established for this study to ensure the safety of trial participants. This DSMB is composed of independent faculty members from the Moi University College of Health Sciences, Aga Khan University Hospital (Kenya), and the MOH, who are not otherwise involved with the project. Membership of the DSMB includes the following expertise: Clinical Cardiology, Clinical Trials, Community-Based Research, Implementation Science, and Ethics. All members are independent and free of any project-related financial interest.

After constitution, the DSMB formulated a charter to guide DSMB operations, a living document that can be reviewed at regular intervals to determine whether any changes in procedure are needed, but cover the areas described below.

# Responsibilities of the DSMB

The DSMB is responsible for safeguarding the interests of study participants, assessing the safety and efficacy of study procedures, and monitoring the overall conduct of the study. The DSMB is an independent group and is required to provide recommendations about starting, continuing, and stopping the study. In addition, the DSMB can be asked to make recommendations, as appropriate, to the NHLBI and/or the appropriate institutional review board (IRB) about:

- Efficacy of the study intervention (DSMB only)
- Benefit/risk ratio of procedures and participant burden
- Selection, recruitment, and retention of participants
- Adherence to protocol requirements
- Completeness, quality, and analysis of measurements
- Amendments to the study protocol and consent forms
- Performance of individual centers and core labs
- Participant safety
- Notification of and referral for abnormal findings

The DSMB will also be expected to coordinate with the TREIN/Hy-TREC consortium coordinating centre for preparing regular DSMB reports.

#### **Organization and Interactions**

Communication between the study staff and DSMB members is primarily through the DSMB administrator (ES). It is expected that study investigators will not communicate with DSMB members about the study directly, except when making presentations or responding to questions at open DSMB meetings. The DSMB ES will provide an unbiased staff interface for the DSMB, especially during executive sessions. The ES is responsible for assuring the accuracy and timely transmission of the final recommendations and DSMB minutes.

# Scheduling, Timing, and Organization of Meetings

The DSMB convened prior to initiation of the trial portion of the study to review the study protocol and give approval of the study trial. They will also convene during the period of trial implementation when interim data analysis is available, and when the final data analysis for the study is available. We will schedule three DSMB meetings a year, with the provision for cancellation should there be nothing to report. The DSMB chair will also decide if additional meetings are required in addition to these minimum meetings. Scheduled analyses will be performed by the study biostatisticians and supplied to the DSMB for review prior to each meeting. If the difference in the primary outcome (change in systolic blood pressure) between any of the intervention arms exceeds the a priori limits defined by the study biostatisticians and the DSMB, the project steering committee has the authority and obligation to consider termination of the study. The DSMB will also receive all Serious Adverse Event (SAE) Reports and may request additional information, as needed. If the DSMB chair deems that an unexpected number of SAEs have been reported they may choose to meet off cycle to assess the events and determine what action should be taken. In addition, on-site monitoring visits from a qualified research monitor (Edwin Sang) will be scheduled quarterly until data quality is deemed acceptable and then will be scheduled six monthly for the remainder of the study.

DSMB meetings are held by teleconference and or video conference as appropriate. The purpose of the first meeting was to review and discuss the DSMB charter, to provide an overview of study activities, to review and make recommendations about the protocol(s), and to determine the frequency of interim analyses and whether data will or will not be masked to identity of randomized groups.

The agenda for DSMB meetings is drafted by the ES. The agenda and meeting materials are distributed to the DSMB at least two weeks in advance of the meeting. Before each meeting, when the agenda is sent out, the Chair asks all DSMB members to state whether they have developed any new conflicts of interest since the last formal annual report to NHLBI. If a new conflict is reported, the Chair and staff determine if the conflict

limits the ability of the DSMB member to participate in the discussion. The DSMB also reviews adverse event data, other safety data, quality and completeness of study data, and enrollment data at each meeting to ensure proper trial conduct. At intervals, as noted above, the DSMB also reviews formal interim analyses of the primary end point.

It is expected that all DSMB members will attend every meeting. However, it is recognized that this may not always be possible. Quorum for voting is considered to be half the number of standing members plus one, that is, 3 members for this proposed DSMB. The DSMB may however wish to decide if particular expertise is needed within the quorum for the meeting to be valid. All standing DSMB members are voting members. The Board may also wish to decide in advance whether ad hoc members can vote.

In the case of the STRENGTHS trial, the decision as to whether to recommend early discontinuation of recruitment should be the responsibility of the DSMB based on all available evidence. Unlike trials where toxicity or inferiority of efficacy is readily demonstrable, the STRENGTHS trial is not expected to be stopped early. Safety and efficacy boundaries, however, have been created for the rare situation of unexpected benefit or harm.

#### **Discussion of Confidential Material**

DSMB meetings and calls are organized into open, closed, and executive sessions.

- During the open sessions, information is presented to the DSMB by the STRENGTHS study investigators and NHLBI staff (as appropriate), with time for discussion.
- During the closed sessions, the DSMB and NHLBI program staff will discuss confidential data from the study, including information on efficacy and safety by treatment arm. If the closed session occurs on a conference call, steps will be taken to ensure that only the appropriate participants are on the call, and to invite others to re-join the call only at the conclusion of the closed session.
- The DSMB may elect to hold an executive session in which only the DSMB members and NHLBI Program staff are present in order to discuss study issues independently. Voting on recommendations will follow Roberts' Rules of Order (Robert's Rules of Order Newly Revised (11th Edition) RONR by Henry M. Robert III, William J. Evans (Editor), Daniel H. Honemann (Editor), Thomas J. Balch (Editor), Sarah Corbin Robert, Henry M. Robert III, General Henry M. Robert). If the executive session occurs on a conference call, steps will be taken to ensure that only the appropriate participants are on the call, and to invite others to re-join the call only at the conclusion of the executive session.

At the conclusion of the closed and executive sessions, the participants will be re-convened at the discretion of the Chair, so that the DSMB Chair can provide a summary of the DSMB's recommendations. This provides an opportunity for study investigators, the STRENGTHS DCC, and NHLBI to ask questions to clarify the recommendations before adjournment. Alternatively, the DMSB's recommendations will be communicated by the Chair to the Study PI after the meeting, at the discretion of the Chair.

#### **Reports of DSMB Deliberations**

**Rapid Communication**: The DSMB Secretary will convey to the PI, and the NHLBI staff the immediate outcome of the DSMB meeting in regards to continuation of the study within 24 hours via personal communication, telephone or email.

**Formal minutes**: The DSMB Chair is responsible for the accuracy and transmission of the formal DSMB minutes within 14 days of each meeting or call. These minutes will summarize the key points of the discussion and debate, requests for additional information, response of the investigators to previous recommendations, and the recommendations from the current meeting. The DSMB Chair may sign the minutes or indicate approval electronically via email. Then, the minutes are sent to the Principal investigator, who will be responsible for sending the document to all relevant institutional review boards, the consortium coordinating centre, and the NHLBI program and clinical trials staff. Subsequently, recommendations of the

Board are sent to the STRENGTHS primary study investigator(s); and included in the materials for the subsequent DSMB meeting to be approved by voice vote at that meeting. Once they have been voted and approved by the Board, they will be considered final.

#### Reports to the DSMB

For each meeting, the ES will prepare summary reports to facilitate the oversight role of the DSMB. The DSMB should discuss at the first or subsequent meetings what data they wish to review and how it should be presented.

#### **Statistical Monitoring Guidelines**

At the first meeting, review of the protocol will include review of the statistical analysis plan. The DSMB should discuss the adequacy of that plan. The final plan, whether part of a research protocol or separate document, will be maintained as an appendix in the formulated DSMB charter. The DSMB should discuss the statistical monitoring procedures they propose to follow, in order to guide their recommendations about termination or continuation of the trial. These procedures could include guidelines for early termination for benefit, termination for futility, and termination for safety reasons.

#### **Protocol Violations and Protocol Deviations**

Protocol deviations are accidental or unintentional changes to, or non-compliance with the research study protocol that does not increase risk or decrease benefit; or does not have a significant effect on the subject's rights, safety or welfare; and/or on the integrity of the data. Deviations may result from the action of the subject, researcher, or research staff. Protocol violations on the other hand are accidental or unintentional changes to, or non-compliance with the IREC-approved protocol without prior sponsor and IREC approval. Violations generally increase risk or decrease benefit, affects the subject's rights, safety, or welfare, or the integrity of the data. In the event of a protocol deviation/violation, the PI or designee will report it to NHLBI, IREC and the DSMB as soon as possible after becoming aware, but no later than seven (7) days for protocol violations and 15 days for protocol deviations, including a 'Corrective Action Plan' for review. In addition, the RC will add the protocol deviation/violation to a log of all protocol deviations/violations, which will be maintained in the regulatory binder (Appendix 5).

#### Safety and Efficacy Boundaries

The DSMB should plan to conduct one major interim analysis at approximately 15 months after initiation of recruitment; the exact time being at the DSMB Chair's discretion. This is to allow for sufficient accrual of primary outcome data for a meaningful number of study participants to reasonably assess safety and efficacy of the intervention. This review will not only look at the usual safety data, but will specifically review the hypertension data in light of clinical events such as strokes, myocardial infarctions and deaths.

If an unexpectedly favorable mean change in blood pressure is noted, defined as a decrease of ≥30 mm Hg, this will be considered an unequivocal sign of benefit, and the DSMB may consider advising stopping the study for overwhelming benefit. This decision will also take into account the data regarding clinical events, especially mortality.

If an unexpectedly unfavorable mean change in blood pressure is noted, defined as an increase of ≥20 mm Hg, this will be considered as an unequivocal sign of harm and the DSMB may consider advising stopping the study for overwhelming harm. This decision will also take into account the data regarding clinical events, especially mortality.

There are no futility boundaries being set for this study given the short/intermediate term follow-up.

Should the DSMB recommend early stopping or modification of the protocol the following steps will be undertaken:

- A meeting will be held between the Principal Investigator and the DSMB to discuss the issues.
- The Principal Investigator will call a meeting with the Steering Committee, as well as the NHLBI program staff representatives. Discussions should be limited to blinded data whenever possible. This discussion should result in agreed actions based on DSMB recommendations.

#### **Ethical Approval**

The protocol for this study, data collection tools, and any subsequent amendments will receive approval from the Moi/MTRH IREC.

#### 12. Team Roster

Table 2: STRENGTHS Team Roster

| Name | Role |
|--------------------------|---------------------|
| Dr. Constantine Akwanalo | PI |
| Dr. Jemima Kamano | Co-PI |
| Josephine Andesia Kisato | Project coordinator |
| Dr. Benson Njuguna | Co-investigator |
| Prof. Violet Naanyu | Co-investigator |
| Dr. Ann Mwangi | Co-investigator |
| Dr. Timothy Mercer | Co-investigator |
| Dr. Rajesh Vedanthan | Co-investigator |
| Dr. Sonak Pastakia | Co-investigator |
| Dr. Jonathan Dick | Co-investigator |
| Dr. Makeda Williams | Co-investigator |
| Dr. Gerald Bloomfield | Consultant |
| Tom Valente | Consultant |
| Eric Finkelstein | Consultant |
| Juliet Miheso | Research Assistant |
| Agneta Pkassan | Research Assistant |
| Eunice Njoki | Research Assistant |
| Monica Nyambura | Data Manager |
| Esther Matini Lotokho | Research Assistant |
| Florence Kiwunja Njulu | Research Assistant |
| Godfrey Kutwa | Research Assistant |
| Sally Asere Ekirapa | Research Assistant |

# Policy on oral or written presentation of results

A written policy guiding oral or written presentation of results will be developed.

#### 13. Timeline

Table 3: Planned Enrollment by Sex

| Targeted/Planned Enrollment | | |
|-----------------------------|---------|-------|
| Males | Females | Total |
| 990 | 660 | 1650 |

| | 100 | YEA | AR 1 | 9 9 | YEAR 2 | | | YEAR 3 | | | | YEAR 4 | | | | YEAR 5 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 01 02 03 04 01 02 03 04 | | | 04 | Q2 | 02 | Q4 | 04 | Q2 | 02 | 04 | 4 Q1 Q2 Q3 | | | | | | | | |
| Preparatory Phase | Q. | I UZ | ų3 | Q4 | Q1 | u2 | ų, | Q4 | Q. | U/2 | ų3 | Q4 | Q1 | Ų2 | u <sub>3</sub> | Q4 | Ψī | U/Z | us. | 100 |
| Finalize protocol manuals | | | | | | | | | П | | | | | | | | $\overline{}$ | | $\Box$ | Г |
| Finalize standard operating procedures | | | | | г | | - | | г | | | | - | | | | | $\vdash$ | | T |
| Develop data collection tools | | | | | Г | - | | 4 9 | г | - | 7 92 | | | | 2 18 | | | | 2 15 | T |
| Hire and train staff | | | 4 1 | - 2 | | 0.00 | | 8 9 | | 12 0 | 0.00 | | 0 3 | | 8 3 | | 3 3 | | 8 3 | Г |
| Aim 1 | | | | | | | | | | | | | | | | | | | | _ |
| Observational process mapping and gap assessment | | | | | | | | | | | 200 | | | | S 10 | | | | s | Г |
| Mabaraza | | | | | | | $\vdash$ | | г | | | | | | | | | $\vdash$ | | T |
| Focus Group Discussions | | | | | | | | | | | | | | | | | | | | Г |
| Key Informant Interviews | 8 | | | | | 1 13 | | 1 3 | | Ø ( | 8 | | 1 | | 1 12 | | 3 3 | | 1 12 | Г |
| Baseline network analysis | | | | | | | | 5 0 | Г | 355 | s 300 | | 9 12 | | S 12 | | | | 5 18 | Г |
| Analysis | | | | | | | | | Г | | | | | | | | | | | Γ |
| Sub-Aim 1.1 | | | | | | | | | | | | | | | | | | | | Т |
| Development | | | | | | | | | | 7 | | | | | | | | | - | Γ |
| Acceptability and Feasibility Testing | 8 | | 8 8 | 8 | | 6 8 | | | | 8 | 8 8 | | 8 | | 1 3 | | 8 8 | | 1 3 | Г |
| Aim 2 | | | | | | | | | | | | | | | | | | | | |
| Training of Peers and Clinicians | _ | 1 | | | Г | | | | | | | | | | | | | | s 15 | Г |
| Enrollment | | | | | | | | | | | | | | | | | | | | T |
| Follow-up | | | - | | | | | | | | | | | | | | | | | Г |
| Data Collection | 8 | | 8 8 | 8 | | 8 | | | | | | | | | | | 8 8 | | į į | Γ |
| Data quality audit | | | 305 3 | | Г | 2 30 | | | | 88 | | | | | | | | | | Г |
| Analysis | | | | | | | | | | | | | | | | | | | | |
| Sub-Aim 2.1 | | | | | | | | | | | | | | | | | | | | Т |
| Data collection | | | | | Г | | | | Г | 7 | | | | | | | | | - | Γ |
| Data quality audit | 8 | 9 | 8 8 | 8 | | 8 | | \$ 3 | | 8 | 8 8 | | 1 10 | | 1 18 | | | | į į | Г |
| Analysis | | 0.0 | 20 0 | 0 8 | | 0 0 | | | | 00 0 | 0 25 | | 5 - 35 | | 35 - 30 | | 9 8 | | | |
| Sub-Aim 2.2 | | | 300 3 | | | | | | 99 | | | | | | | | | | | Ξ |
| Data collection | | | | | Г | | | | | | | | | | | | | | | Г |
| Data quality audit | | | | | | | | | | | | | | | | | | | | Г |
| Analysis | 88 | | 88 8 | 8 | | 8 | | å B | | | | | | | | | 1 | | 1 | Г |
| Aim 3 | | | | | | | | | | | | | | | | | | | | |
| Data collection | | | 200 | | | | | | | | | | | | | | | | S 12 | Г |
| Data quality audit | | | | | Г | | | | | | | | | | | | | | | Γ |
| Analysis | | | | | Г | | | | | | | | | | | | | | | |
| Research Products | | | | - | | | | - | | | | | | | | | | | | |
| Community dialogue and input | | * | 15. | * | | * | | * | Г | * | | * | | * | | * | | * | | Г |
| International Advisory Committee Meetings | 100 | × | ii i | × | | × | | × | | × | 9 8 | x | 8 8 | ж | 8 3 | × | 8 3 | × | 8 8 | T |
| International conferences | | 5 | | | | 5 | | - | | 5 | | | | 5 | | <u> </u> | | 5 | 4 6 | T |
| Publications | | 1 | | | <del>-</del> | - | + | | _ | 3 | # | | | , | + | $\vdash$ | | 3 | + | t |

Figure 5: Timeline for overall STRENGTHS Study

#### 14. References

- 1. Forouzanfar MH, Alexander L, Anderson HR, et al. Global, regional, and national comparative risk assessment of 79 behavioural, environmental and occupational, and metabolic risks or clusters of risks in 188 countries, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet (London, England) 2015;386:2287-323.
- 2. Lim SS, Vos T, Flaxman AD, et al. A comparative risk assessment of burden of disease and injury attributable to 67 risk factors and risk factor clusters in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet (London, England) 2012;380:2224-60.
- 3. Mills KT, Bundy JD, Kelly TN, et al. Global Disparities of Hypertension Prevalence and Control: A Systematic Analysis of Population-Based Studies From 90 Countries. Circulation 2016;134:441-50.
- 4. Kenya STEPwise survey for non-communicable diseases risk factors 2015 report: Ministry of Health Kenya Nation Bureau of Statistics

World Health Organisation; 2015.

- 5. Chow CK, Teo KK, Rangarajan S, et al. Prevalence, awareness, treatment, and control of hypertension in rural and urban communities in high-, middle-, and low-income countries. JAMA: the journal of the American Medical Association 2013;310:959-68.
- 6. Irazola VE, Gutierrez L, Bloomfield G, et al. Hypertension Prevalence, Awareness, Treatment, and Control in Selected LMIC Communities. Global Heart;11:47-59.
- 7. Dale J, Caramlau IO, Lindenmeyer A, Williams SM. Peer support telephone calls for improving health. The Cochrane database of systematic reviews 2008:Cd006903.
- 8. The State of the Health Referral System in Kenya: Results from a Baseline Study on the Functionality of the Health Referral System in Eight Counties. Ministry of Health. 2013.
- 9. Ilboudo TP, Chou YJ, Huang N. Compliance with referral for curative care in rural Burkina Faso. Health policy and planning 2012;27:256-64.
- 10. Uwemedimo OT, Arpadi SM, Chhagan MK, et al. Compliance with referrals for non-acute child health conditions: evidence from the longitudinal ASENZE study in KwaZulu Natal, South Africa. BMC health services research 2014;14:242.
- 11. Kallander K, Tomson G, Nsungwa-Sabiiti J, Senyonjo Y, Pariyo G, Peterson S. Community referral in home management of malaria in western Uganda: a case series study. BMC international health and human rights 2006;6:2.
- 12. WHO. World Health Report 2000, health systems: improving performance: Geneva: World Health Organization.; 2000.
- 13. Murray SF, Pearson SC. Maternity referral systems in developing countries: current knowledge and future research needs. Social science & medicine (1982) 2006;62:2205-15.
- 14. Josyula S, Taylor KK, Murphy BM, Rodas D, Kamath-Rayne BD. Obstetric referrals from a rural clinic to a community hospital in Honduras. Midwifery 2015;31:1054-9.
- 15. Brennan AT, Long L, Maskew M, et al. Outcomes of stable HIV-positive patients down-referred from a doctor-managed antiretroviral therapy clinic to a nurse-managed primary health clinic for monitoring and treatment. AIDS (London, England) 2011;25:2027-36.
- 16. UNICEF. Towards universal access: scaling up priority HIV/AIDS interventions in the health sector. Progress Report 2009. Towards universal access: scaling up priority HIV/AIDS interventions in the health sector Progress report 2009: OMS; 2009.
- 17. Levitt NS, Puoane T, Denman CA, et al. Referral outcomes of individuals identified at high risk of cardiovascular disease by community health workers in Bangladesh, Guatemala, Mexico, and South Africa. Global health action 2015;8:26318.
- 18. Backman G, Hunt P, Khosla R, et al. Health systems and the right to health: an assessment of 194 countries. The Lancet;372:2047-85.
- 19. Levitt NS, Puoane T, Denman CA, et al. Referral outcomes of individuals identified at high risk of cardiovascular disease by community health workers in Bangladesh, Guatemala, Mexico, and South Africa. Global health action 2015;8.
- 20. Kowalewski M, Jahn A, Kimatta SS. Why do at-risk mothers fail to reach referral level? Barriers beyond distance and cost. African journal of reproductive health 2000;4:100-9.

- 21. Pembe AB, Urassa DP, Darj E, Carlsted A, Olsson P. Qualitative study on maternal referrals in rural Tanzania: decision making and acceptance of referral advice. African journal of reproductive health 2008;12:120-31.
- 22. Pembe AB, Carlstedt A, Urassa DP, Lindmark G, Nystrom L, Darj E. Effectiveness of maternal referral system in a rural setting: a case study from Rufiji district, Tanzania. BMC health services research 2010;10:326.
- 23. Bahous MC, Shadmi E. Health information exchange and information gaps in referrals to a pediatric emergency department. International journal of medical informatics 2016;87:68-74.
- 24. Orimadegun AE, Akinbami FO, Akinsola AK, Okereke JO. Contents of referral letters to the children emergency unit of a teaching hospital, southwest of Nigeria. Pediatric emergency care 2008;24:153-6.
- 25. Funnell MM. Peer-based behavioural strategies to improve chronic disease self-management and clinical outcomes: evidence, logistics, evaluation considerations and needs for future research. Family Practice 2010;27:i17-22.
- 26. Chang LW, Kagaayi J, Nakigozi G, et al. Effect of peer health workers on AIDS care in Rakai, Uganda: a cluster-randomized trial. PloS one 2010;5:e10923.
- 27. Deering KN, Shannon K, Sinclair H, Parsad D, Gilbert E, Tyndall MW. Piloting a peer-driven intervention model to increase access and adherence to antiretroviral therapy and HIV care among street-entrenched HIV-positive women in Vancouver. AIDS patient care and STDs 2009;23:603-9.
- 28. Gusdal AK, Obua C, Andualem T, Wahlstrom R, Chalker J, Fochsen G. Peer counselors' role in supporting patients' adherence to ART in Ethiopia and Uganda. AIDS care 2011;23:657-62.
- 29. Medley A, Kennedy C, O'Reilly K, Sweat M. Effectiveness of peer education interventions for HIV prevention in developing countries: a systematic review and meta-analysis. AIDS education and prevention: official publication of the International Society for AIDS Education 2009;21:181-206.
- 30. Wu CJ, Chang AM, Courtney M, Kostner K. Peer supporters for cardiac patients with diabetes: a randomized controlled trial. International nursing review 2012;59:345-52.
- 31. Funnell MM. Peer-based behavioural strategies to improve chronic disease self-management and clinical outcomes: evidence, logistics, evaluation considerations and needs for future research. Family practice 2010;27 Suppl 1:i17-22.
- 32. Smith SM, Paul G, Kelly A, Whitford DL, O'Shea E, O'Dowd T. Peer support for patients with type 2 diabetes: cluster randomised controlled trial. BMJ (Clinical research ed) 2011;342:d715.
- 33. Cabassa LJ, Camacho D, Velez-Grau CM, Stefancic A. Peer-based health interventions for people with serious mental illness: A systematic literature review. Journal of psychiatric research 2016;84:80-9.
- 34. Hatcher AM, Turan JM, Leslie HH, et al. Predictors of linkage to care following community-based HIV counseling and testing in rural Kenya. AIDS and behavior 2012;16:1295-307.
- 35. Okeke NL, Ostermann J, Thielman NM. Enhancing linkage and retention in HIV care: a review of interventions for highly resourced and resource-poor settings. Current HIV/AIDS reports 2014;11:376-92.
- 36. Kelly E, Fulginiti A, Pahwa R, Tallen L, Duan L, Brekke JS. A pilot test of a peer navigator intervention for improving the health of individuals with serious mental illness. Community mental health journal 2014;50:435-46.
- 37. Gabitova G, Burke NJ. Improving healthcare empowerment through breast cancer patient navigation: a mixed methods evaluation in a safety-net setting. BMC health services research 2014;14:407.
- 38. Maxwell AE, Jo AM, Crespi CM, Sudan M, Bastani R. Peer navigation improves diagnostic follow-up after breast cancer screening among Korean American women: results of a randomized trial. Cancer causes & control: CCC 2010;21:1931-40.
- 39. Thorogood M, Connor MD, Lewando-Hundt G, Tollman S, Ngoma B. Secondary prevention of strokeresults from the Southern Africa Stroke Prevention Initiative (SASPI) study. Bull World Health Organ 2004;82:503-8.
- 40. Standards of medical care in diabetes--2013. Diabetes care 2013;36 Suppl 1:S11-66.
- 41. Kim JW, Bosworth HB, Voils CI, et al. How well do clinic-based blood pressure measurements agree with the mercury standard? Journal of general internal medicine 2005;20:647-9.

- 42. Nsanzimana S, Ruton H, Lowrance DW, et al. Cell phone-based and internet-based monitoring and evaluation of the National Antiretroviral Treatment Program during rapid scale-up in Rwanda: TRACnet, 2004-2010. Journal of acquired immune deficiency syndromes (1999) 2012;59:e17-23.
- 43. Bloomfield GS, Vedanthan R, Vasudevan L, Kithei A, Were M, Velazquez EJ. Mobile health for non-communicable diseases in Sub-Saharan Africa: a systematic review of the literature and strategic framework for research. Globalization and health 2014;10:49.
- 44. Mamlin BW, Biondich PG, Wolfe BA, et al. Cooking Up An Open Source EMR For Developing Countries: OpenMRS A Recipe For Successful Collaboration. AMIA Annual Symposium Proceedings 2006:2006:529-33.
- 45. Genberg BL, Shangani S, Sabatino K, et al. Improving Engagement in the HIV Care Cascade: A Systematic Review of Interventions Involving People Living with HIV/AIDS as Peers. AIDS and behavior 2016:20:2452-63.
- 46. Raut A, Thapa P, Citrin D, et al. Design and implementation of a patient navigation system in rural Nepal: Improving patient experience in resource-constrained settings. Healthcare (Amsterdam, Netherlands) 2015;3:251-7.
- 47. Hendren S, Fiscella K. Patient navigation improves the care experience for patients with newly diagnosed cancer. Journal of clinical oncology: official journal of the American Society of Clinical Oncology 2014;32:3-4.
- 48. Freeman HP. The origin, evolution, and principles of patient navigation. Cancer epidemiology, biomarkers & prevention: a publication of the American Association for Cancer Research, cosponsored by the American Society of Preventive Oncology 2012;21:1614-7.
- 49. Hopkins J, Mumber MP. Patient navigation through the cancer care continuum: an overview. Journal of oncology practice 2009;5:150-2.
- 50. Fillon M. Can patient navigation help resolve gaps in cancer care? Journal of the National Cancer Institute 2011:103:1815-7.
- 51. Park PH, Wambui CK, Atieno S, et al. Improving Diabetes Management and Cardiovascular Risk Factors Through Peer-Led Self-management Support Groups in Western Kenya. Diabetes care 2015;38:e110-1.
- 52. Rakhi Karwa, Tim Mercer, Mercy Maina, et al. Leveraging HIV peer based support to facilitate healthcare system transitions. UNPUBLISHED.
- 53. Voils CI, Maciejewski ML, Hoyle RH, et al. Initial validation of a self-report measure of the extent of and reasons for medication nonadherence. Medical care 2012;50:1013-9.
- 54. Division Of Non-Communicable Diseases, Ministry Of Health. Kenya National Guidelines For Cardiovascular Diseases Management. 2018
- 55. Naanyu V, Sidle JE, Frankel RM, Ayuku D, Nyandiko WM, Inui TS. Rooting inquiry in tradition: the health baraza as a tool for social research in Kenya. Qualitative health research 2011;21:14-26.
- 56. Collins GS, Altman DG. An independent external validation and evaluation of QRISK cardiovascular risk prediction: a prospective open cohort study. BMJ (Clinical research ed) 2009;339:b2584.
- 57. Kengne AP, Awah PK, Fezeu LL, Sobngwi E, Mbanya JC. Primary health care for hypertension by nurses in rural and urban sub-Saharan Africa. J Clin Hypertens (Greenwich) 2009;11:564-72.
- 58. Mendis S, Johnston SC, Fan W, Oladapo O, Cameron A, Faramawi MF. Cardiovascular risk management and its impact on hypertension control in primary care in low-resource settings: a cluster-randomized trial. Bull World Health Organ 2010;88:412-9.
- 59. He J, Irazola V, Mills KT, et al. Effect of a Community Health Worker-Led Multicomponent Intervention on Blood Pressure Control in Low-Income Patients in Argentina: A Randomized Clinical Trial. JAMA: the journal of the American Medical Association 2017;318:1016-25.
- 60. Ogedegbe G, Plange-Rhule J, Gyamfi J, et al. Health insurance coverage with or without a nurse-led task shifting strategy for hypertension control: A pragmatic cluster randomized trial in Ghana. PLoS medicine 2018;15:e1002561.
- 61. Little RJ, D'Agostino R, Cohen ML, et al. The prevention and treatment of missing data in clinical trials. The New England journal of medicine 2012;367:1355-60.

- 62. Panel on Handling Missing Data in Clinical Trials. The Prevention and Treatment of Missing Data in Clinical Trials. Washington, DC: National Academies Press; 2010.
- 63. Li T, Huftless S, Dickersin K, et al. Minimal standards in the prevention and handling of missing data in observational and experimental patient-centered outcomes research. : Guidance document prepared for Patient Centered Outcomes Research Institute (PCORI); 2012.
- 64. Rubin DB. Multiple Imputation for Nonresponse in Surveys. New York: Wiley & Sons; 2004.
- 65. Daniels MJ, Hogan JW. Missing Data in Longitudinal Studies: Strategies for Bayesian Modeling and Sensitivity Analysis. Boca Raton: Chapman & Hall / CRC Press; 2008.
- 66. Hogan JW, Laird NM. Mixture models for the joint distribution of repeated measures and event times. Statistics in medicine 1997;16:239-57.
- 67. Hogan JW, Roy J, Korkontzelou C. Handling drop-out in longitudinal studies. Statistics in medicine 2004;23:1455-97.

# Appendix 1: Screening for eligibility tool

# STRENGTHS SCREENING/ELIGIBILITY TOOL Inclusion Criteria

| | Questions | Response | Code |
|---|---|---|---|
| QA-1 | Participant ID | Participant ID | |
| QA-2 | Encounter Date | Date of Encounter | Day/Month/Year |
| QA-3 | Name of the Interviewer | Kisato J.<br>Miheso J.<br>Parklea A.<br>Mwangi Njoki E.<br>Njuguna B.<br>Akwanalo C.<br>Kamano J.<br>Vedanthan R.<br>Other. | 1<br>2<br>3<br>4<br>5<br>6<br>7<br>8 |
| QA-4 | Is patient at least 18 years of age or older? | Yes<br>No [Do no continue-ineligible] | |
| QA-5 | Enrolled in AMPATH CDM program with hypertension. | Yes<br>No | 1 2 |

If referred up, confirm (must meet at least one of the following criteria):

| | in referred up, commit (must meet at least one of the following enteria). | | |
|---|---|---|---|
| | Questions | Response | Code |
| QB-1 | Uncontrolled blood pressure (SBP ≥ 140 or DBP ≥ 90) on 3 or more anti-hypertensive medication? | Yes<br>No | 1 0 |
| QB-2 | Have signs or symptoms of end-organ damage (dyspnoea on exertion, leg edema, reduced urine output, focal weakness) | Yes<br>No [Go to QB-4] | 1 0 |
| QB-3 | [If QB-2=1] Please state the sign(s) or symptom(s) of endorgan damage (check all that apply): | Dyspnea on Exertion<br>Leg Edema<br>Reduced Urine Output<br>Focal Weakness | 2 3 |
| QB-4 | Have suspected secondary causes of hypertension (age <35 years, HIV, or | Yes<br>No [Go to QB-6] | |

| | pregnancy)? | | |
|---|---|---|---|
| QB-5 | [If QB-4=1] Please state the suspected secondary causes (check all that apply): | Ag <35 years<br>HIV<br>Pregnancy | 2 |
| QB-6 | Any other concerning condition that the clinician suspects to be attributable to hypertension for which they would seek a higher level of care | Yes<br>No | 1 0 |
| QB-7 | Referral up criteria confirmed (if yes to at least one of the previous questions). | Yes<br>No | 1 0 |

Go to QD-1

If referred down, confirm (must meet at least one of the following criteria):

| | Questions | Response | Code |
|---|---|---|---|
| QC- | Patient has stable,<br>uncomplicated hypertension,<br>defined as controlled BP<br>(SBP <140 and DBP < 90) for<br>3 or more consecutive visits<br>and has no evidence of new<br>end-organ damage | Yes<br>No | 1 0 |
| QC- | The treating clinician recommends care at a lower level | Yes<br>No | 1 0 |
| QC- | If Q2= 0, explain clinician's reason. | Clinician's reason | |
| QC- | Referral down confirmed (if yes to at least one of the questions). | Yes<br>No | 1 0 |

Exclusion Criteria (if patient meets any of the following):

| | Questions | Response | Code |
|---|---|---|---|
| QD- | Patient has an acute illness requiring immediate medical attention? | Yes<br>No | 1 0 |

| QD- | End stage disease? | Yes<br>No | 1<br>0 |
|---|---|---|---|
| QD- | Terminal illness? | Yes<br>No | 1 0 |
| QD- | Inability to provide informed consent (determined by interviewer)? | Yes<br>No | 1 0 |
| QD- | [If QD-4=Yes] Please explain. | Explain | |
| QD-<br>6 | Did the participant answer ALL of the following questions correctly? 1. Who is the current president? 2. Where are we located? | Yes<br>No | 1 0 |
| QD- | Eligible? | Eligible<br>Not Eligible | 1<br>0 |
| QD-<br>8 | Would you be willing to join the STRENGTHS study? | Yes<br>No | 1 0 |
| QD-<br>9 | Please give reason for declining. | Reason Declined | |
| QD-<br>10 | Consent? | Yes<br>No | 1 0 |

# **Appendix 2: Consent Form STRENGTHS**

#### INFORMED CONSENT FOR STRENGTHS TRIAL

| IREC Study ID #: 0001936 | Participant ID #: |
|--------------------------|-------------------|
| Consenting start time: | |

**Principal Investigators:** Constantine Akwanalo and Jemimah Kamano

**Protocol Title:** Strengthening Referral Networks for Management of Hypertension across the Health Systems (STRENGTHS)

#### **Purpose of this Research Study**

The purpose of this study is to find ways to improve success of referrals for hypertension care in rural Kenya. AMPATH and the Kenya Ministry of Health have implemented a referral network for the care of hypertensive patients in this area across different levels (that is, from dispensary, to health center, sub-county, county and national referral hospitals). AMPATH is planning to evaluate the impact of health information technology (health IT) combined with peer support (trained patients with hypertension) on successful referral for hypertension care and control of blood pressure among patients. We therefore plan to compare the impact of the combined intervention (that is, health IT and peer support) on blood pressure control versus the usual standard clinical care. The results of this study are not only designed to improve hypertension care in Kenya, but will also be applicable to the management of other chronic diseases in Kenya and other developing countries.

You are eligible to take part in this research study because you are hypertensive, enrolled in the AMPATH Chronic Disease Management Program and have been referred to another health facility for further care.

# <u>Duration of Participation and Number of People Expected to Participate</u>

<u>Participation Duration:</u> One year <u>Anticipated Number of Subjects:</u> 1600

#### **Description of Procedure**

If you agree to participate in this research study, the following information explains what may be involved.

To evaluate the impact of combining health IT and peer support on the quality of hypertension care, we are dividing the community into two random groups, one with usual clinical care and the other with our referral support intervention (combined health IT with peer support). Depending on the community unit you live in, you might be approached to receive our referral support intervention to help direct your referrals, or have your referral conducted as per the usual care (with no referral support intervention). If you receive the referral support intervention, a peer (patient with hypertension who is trained in supporting other patients with hypertension) will sit with you and clarify any questions you may have about your referral, and provide education and counseling about hypertension. In addition, in planning for your referral visit, the peer will assist you to plan e.g. provide you with information of anticipated costs for the referral, and help with booking an appointment in the facility you've been referred to. On the day of your visit, a different peer stationed at the receiving facility will be waiting to receive you and assist you to navigate through the facility. At the end of your referral visit, the peer will again clarify any questions you may have. Throughout your participation in the study, the peer may call you or even visit you at home to offer you furthur support for your referral.

The clinicians and the services offered will be the same regardless of the community you are coming from. The fees paid, which have been agreed upon by AMPATH and the Ministry of Health, will also remain the same.

At the beginning of the study we will ask you questions concerning your high blood pressure, medications you take, diet, physical activity level and other lifestyle related questions. We will measure your blood pressure and conduct blood tests to measure your lipid ("fat in blood") levels, and how well your kidneys are working using a test called the creatinine test. To do this, we will need to prick you to withdraw blood using a small needle. About 10 mls of blood will be taken and fed into a portable machine that can determine the results of these tests, or transported back to a health facility laboratory for testing. All the blood test results will be immediately made available to you and we will share the results with your clinician. Taken together, the tests conducted will help us determine your risk for future complications of hypertension such as heart disease. We also wish to study the costs and expenses related to your medical care, to see if there is any difference in costs in the two different groups, therefore, we will ask you questions regarding how much you spend for your hypertension care.

We will repeat the above procedures at the end of the one-year period in which you'll be in the study, so that we can see if there has been any change in these results. The one-year results will also be shared immediately with you and your clinician. If we cannot find you at the end of the 1-year period, we will contact you or your relative by phone.

# **Confidentiality of Study Data**

We will not use your name or any other identifying information when we use this information that you are giving us. The only people who will know that you are a research participant are members of the research team who are trained to keep your information confidential and if appropriate, your health care providers and study clinical monitor. No individual identifying information about you will be disclosed to others, except if required by law.

Study records will be stored in locked cabinets in a locked room. Only the study personnel will have access to the information. All computerized information will be protected by access codes known only to the lead researcher and certain designated staff members.

#### **Potential Benefits**

The referral support intervention might lead to more successful referral completion for you, and improved health. In addition, the information gathered during this research study will help AMPATH improve the implementation of this program. You, your family, and your community may therefore benefit from this research.

#### **Potential Risks or Discomforts**

We will only be collecting personal health information that is a routine part of clinical care, as well as the cost information. This information will be shared only with your clinicians, in order to provide you the best clinical care possible.

Risks associated with blood pressure testing are minimal and may include minor pain discomfort, and swelling at the location of the needle prick, small risk of dizziness, light headedness, and fainting. The risk is however no more than what you may experience during your usual routine clinical care visit.

# **Voluntary Participation and Right to Discontinuation**

It is completely voluntary for you to take part in this study. If you choose to take part, you can refuse to answer any question or ask us to stop at any time with no penalty. This will not affect in any manner your ability to receive medical care at any health facility (private/public), or to receive any benefits to which you are otherwise entitled.

# Compensation

Participants will get transport reimbursement at the 6 month and 12 month follow up visit, however, the initial visit, or any costs associated with completing a referral or any usual clinical care will not be provided. A snack will be provided during the consenting and interview procedures as these will take away time from you.

#### **Future Contact**

We would like to follow you up after six and twelve months. We therefore request for your permission to contact you or any other person (if unavailable) as provided in the demographic data form.

#### **Disclosure of Financial Interests**

Funding for conducting this research is provided by the National Institutes of Health, USA, and Grant number: U01HL138636. There are no financial interests to disclose.

#### **Contact Information:**

In case of any questions/complaints regarding this study, please contact: Dr. Constantine Akwanalo
Moi University College of Health Sciences
Eldoret, Kenya
cakwanalo@gmail.com
0722862968

Is it okay for you to participate in this research study?

# 

| NAME OF WITNESS: | |
|----------------------------------------|----------------------------|
| SIGNATURE OF WITNESS: | Date: |
| (Impartial witness) | (Must be dated by witness) |
| NAME OF PERSON OBTAINING CONSENT: _ | |
| SIGNATURE OF PERSON OBTAINING CONSENT: | Date: |
| Consenting stop time: | |

**Appendix 3: Process Evaluation Protocol** 

# STRENGTHS Process Evaluation Protocol

Last Modified: October 9, 2019

#### **Overview of STRENGTHS Process Evaluation**

The purpose of the process evaluation is to identify and correct problems in study implementation during the trial as well as help explain the results of the trial after the fact. The process evaluation for the STRENGTHS project is based on the Saunders framework<sup>1</sup> and will consist of several components: fidelity (quality), dose delivered (completeness), dose received (exposure), dose received (satisfaction), recruitment, reach (participation rate), and context, as demonstrated in the graphic below.

<sup>&</sup>lt;sup>1</sup> Saunders RP, Evans MH, Joshi P. Developing a process-evaluation plan for assessing health promotion program implementation: a how-to guide. *Health Promotion Practice*. 2005; Apr; 6(2): 134-47.


Each process evaluation component will be assessed using several data collection tools. The protocol below goes over each of the individual data collection tools in detail.

A Process Evaluation REDCAP will be utilized for the management of all quantitative data. Data will be entered by research assistants, verified by the research coordinators and data manager, and analyzed by the statistics team. Qualitative data will be transcribed by the research assistants and analyzed by the research coordinators using NVivo software.

# Acronyms:

BP - Blood Pressure

CDM - Chronic Disease Management

FGD – Focus Group Discussions

HIT – Health Information Technology

KII - Key Informant Interviews

PN - Peer Navigators

RA - Research Assistant

SOP – Standard Operating Procedures

UC - Usual Care

STRENGTHS Protocol v 9.0. 2020-09-10

# 1. Fidelity (Quality)

Aim: To assess how well the trial was implemented as planned Specific aims: To assess the fidelity of a) data collection and entry and b) the intervention delivery

# a) Fidelity of Data Collection and Entry:

#### **Data Collection Observation**

#### Participants:

All members of the research staff that will be collecting data from participants will be observed.

#### Methods:

A study investigator and the research coordinator will observe research staff at the beginning of the study or at the point of hiring (for new staff). Additional observation will be conducted at 3 and 12 months if determined to be needed. The principal investigator and research coordinator will be provided with a checklist of expected behaviors and actions and will check off items as they are completed. The checklist items will be based on the study protocol procedures. The checklist will assess:

Measurement taking: BP, height, weight, waist circumference, using point of care machine (fasting blood sugar, lipid profile)

Survey conduct and connection to participant during survey administration (observe each surveyor 3-4 times and give feedback). Includes Costing Questionnaire and Social Network Survey. Informed consent procedure (includes eligibility and consent forms, proper use of REDCap, and study explanation)

# Outcomes and Analysis:

The statistics team will summarize adherence for each checklist item, and each research staff member's score will be calculated as percent completion. The principal investigator and research coordinator will identify problem areas and provide individual feedback and follow-up training as necessary.

#### **Data Entry**

#### Participants:

All members of the research staff that will be entering data from participants at baseline and/or 3 or 12 months will be observed.

#### Methods:

The data manager and research coordinator will ensure that the following data entry checks are being utilized per the Data Management SOP: double data entry of paper forms for critical fields built into the data management system and out of range checks built into the data management system.

#### Outcomes and Analysis:

The data manager and research coordinator will determine the adherence to the Data Management SOP to assess if the double data entry and out of range checks were implemented as intended. Data manager will utilize quality control feature of REDCAP to determine how many validation errors are made per research assistant, as defined in the Data Management SOP.

# b) Fidelity of Intervention Delivery:

# **Field Observation:**

#### Participants:

All PNs and clinicians enrolled in the study will be observed.

#### Methods

Trained research staff will observe PN actions and interactions by month 3 of the intervention during a site visit. The research staff will be provided with a checklist of expected behaviors and actions and will check off actions as they are completed. The checklist items will be based on the PN guides and designed to assess whether or not their role is being implemented as intended. If needed based on performance (on a case-by-case basis based on results reported on the field observation checklist), additional field observation can be conducted subsequently.

Trained research staff will also observe clinician actions and interactions by month 3 of the intervention during a site visit. If needed based on performance, additional field observation can be conducted subsequently. The research staff will be provided with a checklist of expected behaviors and actions and will check off actions as they are completed. The checklist items will be based on the clinician guides and designed to assess whether or not their role is being implemented as intended.

# **Outcomes and Analysis:**

The statistics team will summarize adherence for each checklist item, and each PN's score will be calculated as percent completion. Adherence will be compared by arm (as applicable), age, gender, and geographical region. The research staff will identify problem areas based on items not conducted (as per the field observation checklist) and will provide individual feedback and follow-up training as necessary. Should certain PNs not meet the expectations after additional training, they will be replaced with another PN from the same community unit.

# **Written Test:**

#### Participants:

Every PN will be given written tests.

#### Methods:

Separate written tests will be given to the PNs assessing knowledge of hypertension care, understanding of the referral system, as well as psychosocial support and patient communication

The test will be translated into Kiswahili and will be administered at baseline (following training) and 6 months.

# **Outcomes and Analysis:**

The statistics team will summarize the results from the written test and do comparisons by groups (geographical region, age, gender, and intervention arm). PN ID numbers will be recorded on the test form to link the baseline and follow-up tests. Each PN's score will be calculated as percent completion. The research staff will identify problem areas and provide individual feedback and follow-up training as necessary based on preliminary analysis of the baseline test. A score lower than 80% will be flagged for review by the principal investigator and/or the research coordinator, and will be evaluated on a case-by-case basis to determine if additional training/feedback is necessary.

#### **Focus Group Discussions:**

#### Participants:

FGDs will be conducted amongst consenting trial participants who have been retained in the trial, participants who dropped out of the trial (based on the clinical definition of a drop-out as someone who has not returned for care in 3 months since the last scheduled appointment), and among PNs. Two clusters from the intervention arm and two clusters in the UC arm will be randomly selected in which one FGD will

be conducted in each consisting of 8-10 randomly selected participants from the intervention arm (for a total of 4 FGDs). UC participants will be recruited from different health facilities in the applicable cluster.

| Retained Participants | | | Participa<br>droppe | | Peer<br>Navigator | |
|---|---|---|---|---|---|---|
| Cluster 1 | Cluster 2 | Cluster 3 | Cluster 4 | All Clusters | All Clusters | All Clusters |
| HIT + peer support | HIT + peer support | UC | UC | HIT + peer<br>support | UC | HIT + peer<br>support |

#### Method:

FGDs will be conducted at approximately 8 months. Data collected through focus group discussions will be used to evaluate fidelity as well as other components of the framework as noted throughout this protocol. A summary of all data collected through FGDs is noted below.

# Participant FGD will:

- Assess participant perceptions of the different intervention components, including the PN and rural clinician activities
- Determine if the intervention is acceptable to participants
- Identify barriers to use and points of successful use of the intervention
- Elicit suggestions from participants about improving the intervention effectiveness

#### PN FGD will:

- Assess if they think peer navigation is helpful for participant care
- Assess perceptions of participant engagement
- Determine if the intervention is acceptable to the providers
- Identify barriers to use and points of successful use of the intervention
- Ascertain if interventions are meeting trial arms and objectives
- Elicit suggestion for improvement

#### **Outcomes and Analysis:**

Content analysis of the FGD data from transcripts of the audio-recordings and notes taken by facilitators during the discussion will be performed using NVivo software. For the participant FGD, the following a priori codes will be used: perceptions of PN and rural physicians, perceptions of intervention activities, importance of hypertension care, importance of referral pathways, and quality of referral services. For the PN FGD, the following a priori codes will be used: perceptions and concerns related to HIT and peer support, cognitive issues around patient interaction (perceived benefit, participant receptivity), emotional elements (frustrations, fears, expectations), and the impact of gender dynamics. Significant inductive (emerging) codes will be identified.

#### Semi-structured interviews with clinicians

#### Participants:

Approximately 18 clinicians will be interviewed at 8 months (at least one from the primary and secondary level from each cluster, and at least 2 from the tertiary level; Moi Teaching and Referral Hospital)

#### Methods:

Trained research staff will conduct semi-structured interviews with the rural clinicians using a structured question guide with the following goals:

- Assess if they think the intervention (use of HIT and peer support) is helpful for participant care
- Determine if the intervention is acceptable to the providers

- Identify barriers to use and points of successful use of the intervention
- Ascertain if interventions are meeting trial arms and objectives
- Elicit suggestion for improvement
- Assess how HIT and peer support impacts patient-clinic interaction

#### **Outcomes and Analysis:**

Content analysis of the interviews from transcripts of the audio-recordings and notes taken by interviewers will be performed using NVivo software. The following a priori codes will be used: perceptions and concerns related to managing the HIT and peer support, cognitive issues around intervention (perceived benefit, participant receptivity), emotional elements (frustrations, fears, expectations), and impact of gender dynamics. Significant inductive (emerging) codes will be identified.

# 2. Dose Delivered (Completeness)

Aim: To determine the number of units of each intervention delivered and if they included the necessary components

Specific aims: To determine if the referral services were provided to participants and in accordance with the components as outlined in the training manuals

# **Participant Self-Reports**

#### Methods:

At the conclusion of 6-month and 12-month visits, 5 randomly selected participants will fill out a brief checklist of tasks completed during the meeting. The checklist will include items assessing PN referral services provided during the visit. These sheets, which will be available in both English and Swahili, will be collected approximately every 3 months when research staff conduct site visits.

#### Outcomes and Analysis:

The statistics team will summarize task completion by individual facility and by arm over the 12 months.

#### 3. Dose Received (Exposure)

*Aim:* To assess to what extent participants were actively engaged with and receptive to the intervention, including initial use and continued use.

Specific aims: To assess participant engagement with the intervention as well as UC, both from the participant and PN perspectives.

# **Focus Group Discussions**

Conducted as outlined in 1. b) III.

## Semi-structured interviews with rural clinicians

Conducted as outlined in 1. b) IV.

#### Field Observation

Conducted as outlined in Section 1. B) I.

#### **Outcomes and Analysis:**

Descriptive statistics will be performed with stratified analysis by relevant demographic characteristics as appropriate.

# 4. Dose Received (Satisfaction)

Aim: To assess the level of participant and provider satisfaction both with the intervention and with their interactions with project staff

Specific aims: To assess the level of participant and provider satisfaction with the implementation of the intervention, as well as UC.

# **Focus Group Discussions**

Conducted as outlined in Section 3a) with focus on participant and provider satisfaction with the intervention components

#### Semi-structured interviews with rural clinicians

Conducted as outlined in Section 3b) with focus on provider satisfaction with the intervention components.

#### 5. Reach (participation rate)

Aim: To determine what percentage of the enrolled participants that participated in the intervention. Specific Aim: To determine the percentage of patients being referred who met with both the PN at their referring facility, as well as the PN at their receiving facility. This will thereby assess retention. Barriers to participation will also be assessed.

#### Clinic Attendance in Usual Care

#### Participants:

Every study participant in the UC arm.

#### Methods:

Every study participant in the UC arm will have their clinical attendance data extracted. Clinic attendance is defined as the completion of a CDM form. The data team will extract dates of CDM clinic attendance from the AMRS for each study participant at 12 months.

# Outcomes and Analysis:

The statistics team will summarize the number of clinic appointments over 12 months by arm.

# **Peer Navigator Encounter in Intervention Arm**

# Participants:

All patient encounter data will also be extracted from the research database for each participant in the intervention. A patient encounter is defined as the completion of a patient encounter form by the PN.

#### Methods:

Every study participant in the intervention arm (receiving HIT and peer support) will also have their encounter data extracted as defined above.

#### **Outcomes and Analysis:**

The statistics team will summarize the number of encounters over 12 months by arm.

#### **Focus Group Discussions**

Conducted as outlined in Section 3a). Specifically, the drop-out focus groups will help assess why certain participants stopped participating.

# 6. Recruitment

*Aim:* To assess what procedures were used to attract participants and what percentage of eligible participants were enrolled out of the total number recorded as eligible during screening.

*Specific Aim:* To determine which enrollment procedures were utilized to screen patients eligible for enrollment, and monitor enrollment procedures.

# Field built into eligibility form

#### Participants:

Research staff involved in enrolling participants will be prompted by the screening and eligibility form on the data management software

#### Methods:

The screening and eligibility form on the project REDCap will prompt research staff to type in a reason when eligible participants choose not to enroll. For patients that do enroll, research staff will indicate which enrollment procedures were utilized. The data management program will also log the attempts to contact and enroll participants and the statuses of these attempts through the scheduling module.

# Outcomes and Analysis:

Reports generated by the data management system will be used to evaluate recruitment strategies and improve as necessary. In order to determine what percentage of eligible participants were enrolled, we will first determine how many participants were eligible from each recruitment pathway. From this, the data team can calculate what percentage of eligible patients were enrolled per pathway and in total.

#### Semi-structured interviews with research staff

#### Participants:

Key members of the research staff in Kenya who were most directly responsible for STRENGTHS participant recruitment will be interviewed at 6 months.

#### Methods:

Trained research staff who were not directly involved with participant recruitment will conduct semistructured interviews with the research staff responsible for recruitment using a structured question guide with the following goals:

- Determine what planned and actual recruitment procedures were used to recruit participants
- Identify barriers in recruitment and successful strategies

#### Outcomes and Analysis:

A content analysis of the interviews from transcripts of the audio-recordings and notes taken by interviewers will be performed using NVivo software. The following a priori codes will be used: recruitment procedures, barriers in recruitment, successful recruitment strategies. Significant inductive (emerging) codes will be identified.

## 7. Context

Aim: To assess the aspects of the environment that may influence intervention implementation or study outcomes, including contamination or the extent to which the control group was exposed to the program. Specific aim: To assess the barriers and facilitators to the two intervention arms, from the participant, provider, and staff perspectives

# a) Focus Group Discussions:

Conducted as outlined in Section 3a) with focus on barriers and facilitators to implementing the intervention.

# b) Semi-structured interviews with clinicians and research staff:

| Conducted as outlined in Section intervention. | ns 3b) and 6b) with f | ocus on barriers and | d facilitators to imple | ementing the |
|---|---|---|---|---|

# Appendix 4: Adverse Event and Serious Adverse Event Reporting Form

# STRENGTHS ADVERSE EVENT AND SERIOUS ADVERSE EVENT REPORTING

NOTE: Complete this report within 24 hours of knowledge of an adverse event occurring or worsening after consent. This report must be filled together/reviewed by the principal investigator or delegated co-investigator. All SAEs will require expedited reporting by the PI to the study's DSMB, IREC/IRB, and NHLBI. An expedited report of an SAE will be submitted by email and must be reported to the DSMB, IREC/IRB and the NHLBI within 24 hours of the event being reported to the Investigator. The expedited report will be followed by a detailed, written AE/SAE report as soon as possible.

# **Causal Relationship**

The assessment of the causal relationship is a clinical decision based on all available information at the time of the completion of the CRF. The assessment is based on whether there was a "reasonable causal relationship" to the study interventions. An assessment of "No" would include the existence of a clear alternative explanation or non-plausibility. An assessment of "Yes" indicates that there is a reasonable suspicion that the event is associated with the subject's participation in the study. Factors to be considered in assessing the relationship of the event to study treatment include:

- The temporal sequence from study intervention procedures: The event should occur after the intervention is delivered. The length of time from exposure to event should be evaluated in the clinical context of the event
- Recovery on intervention discontinuation, recurrence on intervention re-introduction:
   Participant's response after discontinuation should be considered in the view of the usual clinical course of the event in question
- Underlying, concomitant, intercurrent diseases: Each event should be evaluated in the context of the natural history and course of the disease being treated and any other disease the participant may have
- Concomitant medication or treatment: Drugs the participant is taking or the treatment the participant receives should be examined to determine whether any of them may be suspected to cause the event in question

# **Alternative possible explanations**

- Concomitant disease: any illness participant has at time of entering the study, excluding the indication for study intervention
- Concomitant drug: any medication the participant was receiving at time of event onset
- Intercurrent disease: any illness the participant may develop during the study
- Underlying disease: the indication the intervention is being tested for

# **SECTION A – INTRODUCTION**

| | Question | Response | Code |
|---|---|---|---|
| QA-1 | Participant ID | Participant ID | |
| QA-2 | Start Date of Event | Start Date<br>Don't Know | //<br>Day/Month/Year |
| | | Stop Date | // |
| | | • | Day/Month/Year |
| QA-3 | End Date of Event | Ongoing | 88 |
| | | Don't Know | 99 |
| QA-3 | Date and time investigator became aware of this event | Date | //<br>Day/Month/Year |
| | became aware or tims event | Time (in 12-hr clock) | <br>hr—min. pm/am |
| | | Results in death | 1 |
| | | Is life threatening | 2 3 |
| | Does this event associated | Results in hospitalisation or prolongation of hospitalisation | 3 |
| 04.4 | with any of the following | Results in persistent or significant | 4 |
| QA-4 | seriousness criteria? (Select | disability or capacity | |
| | all that are appropriate) | (If any of the above are selected, <b>Go to section B</b> ) | |
| | | None of the above ( <b>Go to section c</b> ) | 5 |

# SECTION B - SERIOUS ADVERSE EVENT

| 0_0 | UN B - SERIOUS ADVERSE EVENT | | |
|---|---|---|---|
| | Question | Response | Code |
| QB-1 | Serious Adverse Event, please fill out the details of the event and give specific diagnosis if possible e.g. heart failure, death etc | | |
| QB-2 | What was the <u>intensity</u> of the SAE | Mild (transient in nature and not interfering with normal activities) No [Sufficiently discomforting to interfere with normal activities] Severe [prevents normal activities] Don't know | 1<br>2<br>3<br>99 |
| QB-3 | Is there a reasonable causal relationship to any of the study interventions? (see definitions on page 1) | Yes<br>No | 1 2 |
| QB-4 | What action was taken with the study intervention? | Study intervention withdrawn (Go to QB-5) Study intervention temporary interrupted (Go to QB-5) No action (Go to QB-7) | 1<br>2<br>3 |
| QB-5 | Did event disappear after stopping study interventions? | Yes<br>No<br>Unknown | 1<br>2<br>99 |
| QB-6 | Did event reappear after reintroducing study interventions? | Yes<br>No<br>Study interventions not reintroduced<br>Unknown | 1<br>2<br>3<br>99 |
| QB-7 | Are there any alternative possible explanations for this event? (see definitions on page 1) | Concomitant disease<br>Concomitant drug<br>Intercurrent disease<br>Underlying disease<br>Unknown | 1<br>2<br>3<br>4<br>99 |
| QB-8 | What was the outcome of this event? | Recovered/Resolved Not Recovered/Not Resolved Recovering/Resolving Fatal Recovered/resolved with sequelae Unknown | 1<br>2<br>3<br>4<br>5<br>99 |

# SECTION C - NON-SERIOUS ADVERSE EVENT

| Ques |
|------|
|------|

| QC-1 | Non-Serious Adverse Event, please fill out<br>the details of the event and give specific<br>diagnosis if possible e.g. heart failure, death<br>etc | | |
|---|---|---|---|
| QC-2 | What was the <u>intensity</u> of the non-serious AE | Mild (transient in nature and not interfering with normal activities) No [Sufficiently discomforting to interfere with normal activities] Severe [prevents normal activities] Don't know | 1<br>2<br>3<br>99 |
| QC-3 | Is there a reasonable causal relationship to any of the study interventions? (see definitions on page 1) | Yes<br>No | 1 2 |
| QC-4 | What action was taken with the study intervention? | Study intervention withdrawn (Go to QC-5) Study intervention temporary interrupted (Go to QC-5) No action (Go to QC-7) | 1<br>2<br>3 |
| QC-5 | Did event disappear after stopping study interventions? | Yes<br>No<br>Unknown | 1<br>2<br>99 |
| QC-6 | Did event reappear after reintroducing study interventions? | Yes<br>No<br>Study interventions not reintroduced<br>Unknown | 1<br>2<br>3<br>99 |
| QC-7 | Are there any alternative possible explanations for this event? (see definitions on page 1) | Concomitant disease<br>Concomitant drug<br>Intercurrent disease<br>Underlying disease<br>Unknown | 1<br>2<br>3<br>4<br>99 |
| QC-8 | What was the outcome of this event? | Recovered/Resolved<br>Not Recovered/Not Resolved<br>Recovering/Resolving<br>Recovered/resolved with sequelae<br>Unknown | 1<br>2<br>3<br>4<br>99 |

# **SECTION D - CONCLUSION**

| | Question | Response | Code |
|---|---|---|---|
| QD-1 | Name of the Interviewer/Research Assistant | | |
| QD-2 | Date of documentation | | //<br>Day/Month/Year |
| QD-3 | Name of the Investigator reviewing this information | | |
| QD-4 | Date of Investigator review | | //<br>Day/Month/Year |

# **Appendix 5: Protocol Deviation/Violation Log**

# **Protocol Deviation/Violation Log**

| Description of Protocol Deviation: | Deviation<br>Category* | Deviation<br>Code** | Date Deviation<br>Occurred:<br>(dd/mm/yyyy) | Date IREC/<br>IRB<br>Notified | Principal<br>Investigator's<br>Signature | Date Signed<br>(dd/mm/yyyy) |
|---|---|---|---|---|---|---|

#### \*DEVIATION CATEGORIES:

- A. Safety
- B. Informed Consent
- C. Eligibility
- D. Protocol implementation
- E. Other, specify in log
- \*\*DEVIATION CODES: Numbers listed by the sample protocol deviations

#### Safety (Category A)

- 1. Not reporting an SAE within 24 hours
- 2. Laboratory tests not done
- 3. AE/SAE is not reported to IRB
- 4. Other, specify in log

# Informed Consent (Category B)

- 5. Failure to obtain informed consent
- 6. Consent form used was not current IRBapproved version
- Consent form does not include updates or information required by IRB
- 8. Consent form missing

- 9. Consent form not signed and dated by participant
- Consent form does not contain all required signatures
- 11. Other, specify in log

# Eligibility (Category C)

- 12. Participant did not meet eligibility criterion
- 13. Randomization of an ineligible participant
- 14. Participant randomized prior to completing Baseline Assessment, etc.
- 15. Randomization and/or treatment of participant prior to IRB approval of protocol
- 16. Other, specify in log

## Protocol implementation (Category D)

- 17. Failure to keep IRB approval up to date
- 18. Participant receives wrong treatment
- 19. Participant seen outside visit window
- 20. Use of unallowable concomitant treatments
- 21. Prescribed dosing outside protocol guidelines
- 22. Missed assessment
- 23. Missed visit
- 24. Other, specify in log